CLINICAL TRIAL: NCT00268554
Title: Enhancement of Postocclusive Reactive Hyperaemia
Brief Title: Enhancement of Postocclusive Reactive Hyperaemia by Dipyridamole
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PORH-dipy
Record Dates: First submitted 2005-12-21; First posted 2005-12-22 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Hyperemia; Hypoxia
Keywords: adenosine; caffeine; dipyridamole
MeSH Terms: conditions — Hyperemia; Hypoxia | interventions — Dipyridamole; Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: dipyridamole
Drug: caffeine

SUMMARY:
The purpose of this study is to determine whether dipyridamole enhances postocclusive reactive hyperaemia by increasing extracellular adenosine concentrations during ischemia and reperfusion. Furthermore we hypothesize that dipyridamole augments postocclusive reactive hyperaemia by increasing adenosine receptor stimulation.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers between 18 and 50 years

Exclusion Criteria:

* none specified

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2005-12; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
forearm blood flow

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Rongen, MD,PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud university Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands